CLINICAL TRIAL: NCT04114656
Title: A Randomized, Double-blind, Placebo-controlled, Three-period Two-treatment Incomplete-block Crossover Study to Investigate the Effects of Intravenous GSK3858279 on a Battery of Evoked Pain Tests in Healthy Participants
Brief Title: Effects of Intravenous GSK3858279 on a Battery of Evoked Pain Tests in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated due to meeting protocol defined futility.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 209973; 2019-002609-23 (EudraCT Number)
Record Dates: First submitted 2019-09-12; First posted 2019-10-03 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-09

CONDITIONS: Pain
Keywords: GSK3858279; Crossover study; Pain assessment; Placebo-controlled; Intravenous
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receiving Placebo (Placebo Comparator): All participants will receive a single dose of placebo in either one or two of the three study periods, as per the randomization schedule.
  Interventions: Drug: Placebo
- Participants receiving GSK3858279 (Experimental): All participants will receive a single dose of GSK3858279 in either one or two of the three study periods, as per the randomization schedule.
  Interventions: Drug: GSK3858279

INTERVENTIONS:
Drug: Placebo — Placebo will be available as intravenous (IV) infusion of normal saline (0.9 percent [%] sodium chloride solution).
  Arms: Participants receiving Placebo
Drug: GSK3858279 — GSK3858279 will be available as IV infusion and the dose level to be administered is 3 milligrams (mg) per kilogram (kg).
  Arms: Participants receiving GSK3858279

SUMMARY:
This study will evaluate the mechanistic basis for the analgesic effects of GSK3858279 in humans by using a battery of experimental pain assessments in healthy participants. This will be placebo-controlled, three-period two-treatment crossover study. In each period, participants will receive either GSK3858279 or placebo in a 1:1 ratio. Only healthy male participants will be enrolled into the study. The duration of the study will be approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 to 50 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs and cardiac monitoring.
* Participants with body weight within 50-100 kg and body mass index (BMI) within the range 18 to 30 kg per meter square (kg/m^2) (inclusive).
* Must be male participants: Participants must agree to the following during the intervention period and for at least 90 days after the last dose of study intervention:

  1. Refrain from donating sperm plus, either
  2. Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or
  3. Must agree to use contraception/barrier as detailed below:

  (i) Agree to use a male condom. (ii) And should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Participants with history or presence of/significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* Personal or family history of cardiomyopathy.
* Abnormal blood pressure as determined by the investigator.
* Symptomatic herpes zoster within 3 months prior to screening.
* Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, and TB testing: a positive (not indeterminate) QuantiFERON-TB Gold test.
* Significant allergies to humanized monoclonal antibodies.
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A [IgA] dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
* Lymphoma, leukemia, or any malignancy. Those who are at risk of deoxyribonucleic acid (DNA) repair diseases or any family history of DNA repair disease.
* Alanine transaminase (ALT) greater than (>)1.5 times upper limit of normal (ULN).
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin less than [<]35%).
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT interval (QTc) >450 msec.
* History of Stevens-Johnson syndrome.
* Known immunodeficiency.
* Participants with an acute, recurrent or chronic infection (for example, osteomyelitis), who have been receiving treatment within three months prior to dosing or individuals with an active infection.
* Previous or current history of excessive bleeding or coagulation disorders.
* Previous history of hypertrophic or keloid scarring.
* Any current, clinically significant, known medical condition in particular any existing conditions that would affect sensitivity to cold (such as atherosclerosis, Raynaud's disease, urticaria, and hypothyroidism) or pain (such as disease that causes pain, hypesthesia, hyperalgesia, allodynia, paraesthesia, neuropathy).
* Participants indicating pain tests intolerable at screening. Participants achieving tolerance at >80% of maximum input intensity for cold pressor and electrical pain tests are to be excluded. If pressure pain test tolerance is >80% of maximum input intensity they may be enrolled as per Principal Investigator (PI) judgement.
* History or presence of post-inflammatory hyperpigmentation. Applicable for the participants in the UVB-Modified Intent-To-Treat (MITT) population only.
* Participants with Fitzpatrick skin type IV, V or VI. Applicable for the participants in the UVB-MITT population only.
* Any of the following on the proposed test area on the back: widespread acne, freckles, tattoos, birthmarks or scarring (investigator discretion may be used to determine if small areas may be avoided in the testing area on the back). Applicable for the participants in the UVB-MITT population only.
* A minimal erythema dose (MED) higher than 355 millijoule per square centimeter (mJ/cm^2) at screening. Applicable for the participants in the UVB-MITT population only.
* Past or intended use of over-the-counter or prescription medication including herbal medications within 7 days prior to screening until after follow-up visit.
* Live vaccine(s) within 1 month prior to screening or plans to receive such vaccines during the study.
* Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) or immunosuppressants within 3 months or 5 half-lives (whichever is longer) prior to dosing.
* Treatment with anti-platelet or anti-coagulant agents within 7 days of dosing.
* Major surgery (as per investigator's judgement) within 3 months prior to dosing.
* Participant has made a blood or plasma donation or has had a comparable blood loss (>450 milliliters [mL]) within the last 3 months prior to the Screening Visit. Blood donation during the study is not permitted.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrollment or past participation in any other clinical study involving an investigational study intervention within the last 3 months, 5-half-lives or twice the duration of the biological product before screening in this current study.
* Presence of Hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention.
* Presence of Hepatitis B core antibody (HbcAb) at screening or within 3 months prior to first dose of study intervention.
* Positive Hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Positive Hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention.
* Abnormal clinically significant echocardiogram at screening, as assessed by the investigator.
* Cardiac troponin T or N-terminal pro-brain natriuretic peptide (NT-proBNP) levels out of normal range at screening.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse.
* Estimated glomerular filtration rate (eGFR) of <90 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) or serum creatinine >1.5 times ULN or urine albumin:creatinine ratio of >300 mg per gram (g) at screening.
* Positive Severe acute respiratory syndrome- Coronavirus-2 (SARS-CoV-2) Polymerase chain reaction (PCR) or rapid antigen test at screening. Participants may be re-screened once they present a negative SARS-CoV-2 PCR or rapid antigen test.
* Participants with known Coronavirus Disease-2019 (COVID-19 positive contacts in the past 14 days.
* Regular alcohol consumption within 6 months prior to the study defined as: an average weekly intake of >21 units for males. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Smoker, smoking history or use of tobacco- or nicotine-containing products (for example, nicotine patches or vaporizing devices) within 6 months prior to screening.
* Sensitivity to heparin or heparin-induced thrombocytopenia.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the effects of GSK3858279 on a battery of evoked pain tests in healthy male participants. This study was terminated due to meeting protocol defined futility.
Pre-assignment Details: A total of 21 healthy male participants were enrolled.
Groups:
- Placebo/GSK3858279 3 mg/kg IV/GSK3858279 3 mg/kg IV: Participants received a single dose of Placebo (normal saline i.e.[0.9 percent {%} sodium chloride]) administered intravenously (IV) in treatment period 1 followed by GSK3858279 3 milligrams per kilogram (mg/kg) administered IV in treatment period 2 followed by GSK3858279 3 mg/kg administered IV in treatment period 3. There was a washout of at least 4 weeks between dosing (i.e. Day 1) in each of the study periods.
- GSK3858279 3 mg/kg IV/Placebo/Placebo: Participants received a single dose of GSK3858279 3 mg/kg administered IV in treatment period 1 followed by Placebo (normal saline [0.9%] sodium chloride) administered IV in treatment period 2 followed by Placebo (normal saline [0.9%] sodium chloride) administered IV in treatment period 3. There was a washout of at least 4 weeks between dosing (i.e. Day 1) in each of the study periods.
Period: Treatment Period1+Washout(Up to 28 Days)
Arm/Group | Placebo/GSK3858279 3 mg/kg IV/GSK3858279 3 mg/kg IV | GSK3858279 3 mg/kg IV/Placebo/Placebo
Started (Discontinuation data were collected until the end of the washout irrespective of whether each participant was in a particular period or began washout. The electronic case report form (eCRF) was not designed to differentiate data collection between treatment periods and washout periods) | 11 | 10
Completed | 9 | 7
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Study closed/terminated | 0 | 2
Not completed — Participant reached protocol defined stopping criteria | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Treatment Period2+Washout(Up to 28 Days)
Arm/Group | Placebo/GSK3858279 3 mg/kg IV/GSK3858279 3 mg/kg IV | GSK3858279 3 mg/kg IV/Placebo/Placebo
Started (Discontinuation data were collected until the end of the washout irrespective of whether each participant was in a particular period or began washout. The electronic case report form (eCRF) was not designed to differentiate data collection between treatment periods and washout periods) | 9 | 7
Completed | 9 | 6
Not Completed | 0 | 1
Not completed — Participant reached protocol defined stopping criteria | 0 | 1
Period: Treatment Period 3 (Up to 28 Days)
Arm/Group | Placebo/GSK3858279 3 mg/kg IV/GSK3858279 3 mg/kg IV | GSK3858279 3 mg/kg IV/Placebo/Placebo
Started | 9 | 6
Completed | 9 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/GSK3858279 3 mg/kg IV/GSK3858279 3 mg/kg IV | GSK3858279 3 mg/kg IV/Placebo/Placebo | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.3 (7.93) | 31.1 (7.71) | 30.1 (7.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - White/Caucasian/European heritage | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Posterior Median Ratio to Baseline of Area Under the Curve (AUC 1-8 Days) in Ultraviolet B (UVB) Heat Pain Detection
Description: Thermal pain tests performed first on normal skin contralateral to site of UVB irradiation then on UVB irradiated skin.A 30*30 millimeter(mm)thermode was placed on participant's back. Initial temperature of thermode was 32 degree Celsius(C)and increased by 0.5 degree C/second until participant indicated painful stimulus(pain detection threshold indicated by pushing a button on hand-held feedback control or when temperature of 50 degree C reached).AUC ratio to Baseline derived from log change from Baseline in temperature versus(vs)time of study period calculated via trapezoidal method &normalized & back transformed(exponential)to get ratio to Baseline. Baseline was mean value of 2 assessments taken before each dosing(Day 1).Posterior Median Ratio to Baseline derived from Bayesian analysis updating prior(non-informative)with information collected from study(likelihood).Data reported as 'Median' refers to 'Posterior Median' and '95% Confidence Interval' refers to '95% Credible Interval'.
Time Frame: Baseline (Day 1) and up to Day 8
Population: UVB modified intent to treat (MITT) Population comprised of participants in the MITT Population who also performed at least one UVB Heat Pain detection PainCart assessment on irradiated skin in at least two study periods. Only those participants with data available at specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Ratio
Groups:
- Placebo: All participants who received at least a single IV dose of Placebo on Day 1 in either Period 1 or Period 2 or Period 3 as per randomization schedule.
- GSK3858279 3 mg/kg IV: All participants who received at least a single IV dose of GSK3858279 3 mg/kg on Day 1 in either Period 1 or Period 2 or Period 3 as per randomization schedule.
Arm/Group | Placebo | GSK3858279 3 mg/kg IV
Number analyzed (Participants) | 12 | 12
Ratio | 1.005 [0.980 to 1.030] | 0.998 [0.976 to 1.021]
Statistical Analysis 1: Comparison: Placebo vs GSK3858279 3 mg/kg IV; Test type: Other; Posterior Ratio to placebo = 0.993, 95% CI 2-sided [0.968 to 1.020] — Treatment comparison ratio of GSK3858279 and placebo using posterior median ratio and 95% credible interval is presented. Analysis was performed using Bayesian Mixed Repeated measures Analysis of Covariance (ANCOVA) model

2. Primary Outcome: Posterior Median Ratio to Baseline of AUC (1-15 Days) in Cold Pressor Time to Intolerable Pain Threshold
Description: Participants put non-dominant hand in water bath at 35+/-0.5 degree C.Blood pressure cuff on upper arm inflated to 20mm of Mercury below resting diastolic pressure. Participants then removed hand & directly placed in similar-size bath(1.0+/-0.5 degree C).Participants indicated increase in pain intensity by moving electronic Visual Analogue scale(eVAS) slider when pain detection threshold was reached(first change in sensation from cold non-painful to painful).When pain tolerance was reached, participants removed their hand& blood pressure cuff was deflated.AUC ratio to Baseline derived from log change from Baseline in time to intolerable pain vs time of study period calculated via trapezoidal method &normalized and back transformed(exponential) to get ratio to Baseline.Baseline was mean value of 2 assessments taken before each dosing(Day 1).Posterior Median Ratio to Baseline derived from Bayesian analysis updating prior(non-informative)with information collected from study(likelihood).
Time Frame: Baseline (Day 1) and up to Day 15
Population: MITT Population comprised of all randomized participants who received at least one dose of study treatment and completed at least one PainCart assessment in at least two study periods. Only those participants with data available at specified time points were analyzed. Data reported as 'Median' refers to 'Posterior Median'& data reported as '95% Confidence Interval' refers to'95% Credible Interval'.
Measure: Median (95% Confidence Interval); unit: Ratio
Arm/Group | Placebo | GSK3858279 3 mg/kg IV
Number analyzed (Participants) | 15 | 15
Ratio | 1.05 [0.96 to 1.15] | 1.05 [0.97 to 1.14]
Statistical Analysis 1: Comparison: Placebo vs GSK3858279 3 mg/kg IV; Test type: Other; Posterior ratio to placebo = 1.00, 95% CI 2-sided [0.89 to 1.12] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Posterior Median Ratio to Baseline of AUC (1-15 Days) in Electrical Pain Tolerance Threshold (Single Stimulus)
Description: Two electrodes were placed on clean (scrubbed) skin overlying left tibial bone 100mm distal from caudal end of patella to detect cutaneous electrical pain. Each stimulus(10-Hertz [Hz] tetanic pulse with duration of 0.2 milliseconds) was controlled by a computer-controlled constant current stimulator.Pain intensity after each stimulation was measured using eVAS,until pain tolerance level was reached,or maximum of 50 milliamper(mA) was reached. AUC ratio to Baseline derived from log change from Baseline in mA versus time of study period calculated via trapezoidal method and normalized and back transformed(exponential)to get ratio to Baseline. Baseline was mean value of 2 assessments taken before dosing(Day 1).Posterior Median Ratio to Baseline derived from Bayesian analysis updating prior (non-informative) with information collected from study(likelihood).Data reported as 'Median' refers to'Posterior Median'and data reported as'95% Confidence Interval' refers to '95% Credible Interval'.
Time Frame: Baseline (Day 1) and up to Day 15
Population: MITT Population. Only those participants with data available at specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Ratio
Arm/Group | Placebo | GSK3858279 3 mg/kg IV
Number analyzed (Participants) | 15 | 15
Ratio | 1.09 [1.01 to 1.17] | 1.07 [1.00 to 1.14]
Statistical Analysis 1: Comparison: Placebo vs GSK3858279 3 mg/kg IV; Test type: Other; Posterior ratio to placebo = 0.98, 95% CI 2-sided [0.91 to 1.05] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs), and non-serious adverse events (non-SAEs) were collected up to 302 days
Description: All-cause mortality, SAEs and non-SAEs were collected for the Safety Population that comprised of all randomized participants who received at least one dose of study treatment. Adverse events were presented treatment-wise.
Arm/Group | Placebo | GSK3858279 3 mg/kg IV
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 10/18 | 12/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | GSK3858279 3 mg/kg IV (N=19)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 1 (1) | 2 (3)
Vaccination site pain (General disorders) | 1 (1) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 1 (1)
Application site warmth (General disorders) | 0 (0) | 1 (1)
Catheter site bruise (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Presyncope (Nervous system disorders) | 1 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Urine output increased (Investigations) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT04114656/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT04114656/SAP_001.pdf